# **Protocol Page**



Clinical and technical feasibility of a ultrasuperparamagnetic nanoparticle iron oxide (USPIO)-enhanced magnetic resonance lymph node imaging 2012-0926

# **Core Protocol Information**

| Short Title | USPIO MRI |
|---|---|
| Study Chair: | Haesun Choi |
| Additional Contact: | Ada Lo<br>Michelle W. Haynes<br>Sujaya Rao |
| Additional Memo Recipients: | Recipients List |
| | <b>OPR Recipients</b> (for OPR use only)<br>None |
| | Study Staff Recipients None |
| Department: | Diagnostic Radiology |
| Phone: | 713-745-4693 |
| Unit: | 1473 |
| Full Title: | Clinical and technical feasibility of a ultrasuperparamagnetic<br>nanoparticle iron oxide (USPIO)-enhanced magnetic resonance lymph<br>node imaging |
| Protocol Type: | Standard Protocol |
| Protocol Phase: | N/A |
| Version Status: | Activated 12/11/2014 |
| Version: | 07 |
| <b>Document Status:</b> | Saved as "Final" |
| Submitted by: | Michelle W. Haynes11/20/2014 10:55:28 AM |
| OPR Action: | Accepted by: Melinda E. Gordon 12/1/2014 10:32:01 AM |

# Which Committee will review this protocol?

The Clinical Research Committee - (CRC)

### **Protocol Body**

# 1.0 Background

The accurate nodal staging at the time of initial presentation or during the surveillance of oncologic patients is important in treatment planning and predicting the clinical outcome. Some of these nodes are not easily accessible for tissue diagnosis. The accuracy of the current imaging techniques detecting metastatic nodal disease are, however, notoriously suboptimal and vary greatly depending on the criteria [1-7].

An ultra-small superparamagnetic nanoparticle iron oxide, Combidex® (ferumoxtran-10), has shown promising results in evaluating the lymph nodes in patients with several different solid tumors and locations [8-14]. One of the largest series from Massachusetts General Hospital has shown about 90% sensitivity and 98% specificity in diagnosing the metastatic pelvic lymph nodes in patients with prostate carcinomas with 41% sensitivity and 98% specificity for the nodes less than 5 mm [14]. Our preliminary work using the Combidex® has shown technical feasibility (unpublished data) (Fig 1). This MR imaging contrast, however, is no longer manufactured. Recently a similar superparamagnetic nanoparticle, Feraheme® (ferumoxytol) has been FDA-approved as an iron replacement product in treatment of the iron deficiency anemia in an injectable solution [15]. These two agents are very similar in their size and pharmacokinetics (Table 1) [15, 16]. Once ferumoxytol is injected, like ferumoxtran-10, the colloids are taken by macrophages in RES system, including the liver, spleen and bone marrow. Once it enters the hepatocyte, it breaks down to release the iron. It reaches the nodes within 1-2 days and stays longer than 7 days [15, 16].

These USPIO particles or macrophages, when they reach the reticular endothelial system, such as liver or lymph nodes, create microscopic field gradients resulting in predominant susceptibility effect and generate local field inhomogeneity promoting dephasing the proton spins and increasing proton relaxation rates, which reduces the tissue T2 values. This results in homogenous and significant decrease in signal intensity (SI) on T2 and T2\*-weighted images on MRI [17-19].



Figure 1. Pre- (a) and 24-hour post (b)-Combidex® enhanced T1-weighted images in a patient with bladder cancer showing normal (arrow)and malignant nodes (circle). Notice the size of nodes is less than 5mm.

Table 1. Comparison of Combidex ® and Feraheme®

| | Combidex® (Ferumoxtran-10) | Feraheme® (Ferumoxytol) |
|---|---|---|
| Particle size | <50 nm | 17-31 nm |
| Amount of iron per vial | 210 mg | 510 mg |
| Volume per vial | 10.5ml | 17ml |
| Amount of iron/ml | 20mg/ml | 30 mg/ml |
| Injection rate | 4ml/min with 100 cc N/S | 1 ml/sec (30 mg/sec) |
| Dose | 2.6 mg of Fe/kg | 510 mg/dose - can be repeated after 3 days of the first dose |

The primary goals of the study are to evaluate 1) if Feraheme-enhanced MRI is capable of producing a diagnostic quality of images (technical feasibility) and 2) if Feraheme-enhanced MRI is capable of identifying malignant node as malignant and benign lymph node as benign, once the MRI is technically optimized (clinical feasibility). This study will be a strong foundation of future investigation of the true value of USPIO-enhanced lymph node imaging in clinical patient care and will open the door to the clinical implementation of a non-invasive lymph node imaging in oncologic patients.

Additional potential benefit of USPIO is dramatic improvement of the vascular enhancement on T1-weighted MR images for a length of time during early vascular phase and the contrast has been suggested to use for MR angiography [20] and dynamic liver imaging [21]. In liver imaging, if the early vascular phase of images can be acquired at the same setting with the MR lymph node imaging (MR-LNI), the additional Gd-enhanced MRI may be eliminated in some patients who require reticular endothelial system of liver or lymph node imaging.

In this study, we will also explore the capability of Feraheme-enhanced MRI in producing a diagnostic quality of early vascular phase imaging of liver (technical feasibility).

# 2.0 Objectives

### Primary Objectives:

- 1. To evaluate if the Feraheme®-enhanced MR-LNI is capable of producing diagnostic quality of images once the imaging parameters, including the scan time, are optimized.
- 2. To evaluate the clinical feasibility of MR-LNI in oncologic patients

#### Exploratory Objectives:

Explore the technical feasibility of Feraheme® use in an early vascular phase of liver imaging

### 3.0 Patient Eligibility

#### Patient Selection

A total of 18 patients (maximum allowable sample size with an available fund) will be enrolled.

#### Inclusion Criteria

- 1) Enrolled at MDACC, Written consent
- 2) Measurable nodes on the recent cross sectional imaging (CT, MRI. US) or suspicous lymph nodes for metastasis
- 3) Requiring tissue diagnosis (FNA, core biopsy, surgical biopsy, surgical resection), or clinical follow-ups for at least 6 months.
- 4) Any and all primary disease sites in the abdomen and pelvis will be allowed

### Exclusion Criteria

- 1. Primary or secondary iron overload
- 2. Lactation or pregnant women with child bearing potential will be excluded
- 3. Contraindications for MRI
- 4. Contraindication or allergy to Feraheme® (based on insert)
- 5. Clinically documented or risk of primary or secondary iron overloading (e.g. History of thalassemia, sickle cell anemia, hereditary hemochromatosis, multiple transfusions with any reason), anemia not caused by iron deficiency
- 6. Age under 18

## 4.0 Study Plan and Methods

# 1. Technical feasibility of Feraheme®-enhanced MR-LNI

- 1. A total of 18 patients will be selected in a consecutive fashion. The patients will be referred by one of the clinical collaborators and screened and consented by a research nurse, PI or radiologist collaborators.
- 2. Based on our previous experience with Combidex® and on-going experience of the investigators at Massachusetts General Hospital (MGH) (unpublished data), we will begin with the similar imaging parameters that were used previously. The imaging parameters will be adjusted as needed to optimize the visualization of the nodes.

[Although this process is unpredictable, it may take about 5-10 patients in initial optimization of the imaging parameters and additional 5-10 patients in identification of an optimum scan time. We expect that there will be an overlap of patients between these 2 processes. When image parameters cannot optimize with the first 10 patients, the study will be terminated.]

- 3. MRI will be acquired prior to the injection of Feraheme® and repeated at approximately 48 hours and 72 hours from the time of injection (scan time). The scan time will be adjusted, as needed.
- 4. Based on the on-going experience of MGH (unpublished data), 6mg of iron/kg (maximum 510mg/dose) will be injected at a rate of 1 ml/sec (30 mg/sec) or slower.
- 5. In those without pathologic correlation, all nodes will be followed clinically for at least 6 months.
- 6. The clinical decision will not be based on the results of the MRI.

# Exploration of USPIO use in liver imaging

- 1. Patients undergoing Abdominal MR-LNI for this trial will be selected for additional imaging for liver on day 1.
- 2. On day 1, additional T1WI will be acquired at arterial, portal venous, and delayed venous phases and 5 minutes, 10min and 30min from the time of injection of Feraheme®. This timing will be modified as needed, depending on our experience of the first couple of patients.
- 3. Quality of aorta enhancement at each time point will be evaluated subjectively as an indicator of adequacy of vascular phase of liver images.

### MRI techniques

All MRI data will be acquired using FDA-approved pulse sequences and radiofrequency coils.

# 1.1 Technical feasibility of Feraheme® -enhanced MR-LNI

Four pulse sequences will be acquired as part of this trial:

- 1) A two dimensional (2D) T2-weighted fast spin-echo (T2W-FSE) sequence,
- 2) a 2D T2\*-weighted gradient-echo (T2\*W- GRE) sequence,
- 3) a 2D T1-weighted gradient-echo (T1W-GRE) sequence, and
- 4) a 3D T1W-GRE sequence.

For each sequence, the section thickness will not exceed 5-mm. The total exam time will not exceed 30 minutes.

The pulse sequence will be modified as needed.

### 1.2 Exploration of USPIO use in liver imaging

GRE T1WI will be acquired at arterial, portal venous, and delayed venous phases, following a routine dynamic technique, and 5 minutes, 10min and 30min from the time of injection following injection of Feraheme. Conventional dynamic technique will be used for imaging parameters.

The scan time will be adjusted as needed.

# 5.0 Data Collection and Analysis

All subjective evaluation will be performed based on a consensus of three radiologists.

### Optimization of the imaging parameters

- 1. Based on our previous experience with Combidex® and on-going experience of Massachusetts General Hospital (MGH) (unpublished data), the image data will be collected at approximately 48 hours and 72 hours after the injection of Feraheme®. The scan time will be adjusted as needed.
- 2. The image quality will be graded subjectively (poor, fair, good).
  - 3. The signal intensity (SI) change of a lymph node between the pre- and post- contrast images will be observed subjectively at each time point. The degree of SI change at each time point, then, will be compared each other subjectively and a time point showing the nodes best (greatest signal loss relative to that on pre-contrast images) will be identified (optimum scan time).
  - 4. In those who undergo biopsy or surgical exploration, pathological status of each evaluated lymph node will be recorded whether they are malignant or benign. In those who do not undergo for the tissue diagnosis, nodes will be followed with routine clinical images (CT or MRI) for at least 6 months. The purpose of this step is to exam the technically optimized Feraheme-enhanced MRI sees the malignant node as malignant and benign nodes as benign by subjective evaluation. A statistical analysis is not applicable at this time.

### Exploration of SPIO-enhanced liver imaging

When images of abdomen are available:

- 1. The overall image quality will be graded subjectively (poor, fair, good).
- 2. The quality of aorta enhancement will be graded subjectively (poor, fair, good).
- 3. Statistical analysis is not applicable at this time.

## 6.0 Adverse Events

# **Drug Information**

Drug Information: Package insert [15]

# Adverse Events

Feraheme® may cause serious hypersensitivity reaction and hypotention. The adverse reactions were reported in ≥1% of Feraheme® treated patients for iron deficiency anemia based on the randomized clinical trials. Diarrhea 4.0%, constipation 2.1% and hypotension 1% are among the most common events [15].

# Managing and Reporting Adverse Events and Allergic Reaction

In the event of allergic type reaction, the patients will be treated in the same manner of allergic reaction occurred by an iodinated contrast following M. D. Anderson Cancer Center standard practice. The drug toxicity will be evaluated according to M. D. Anderson Guidelines (CTC version 4). Reporting of adverse events will be according to M. D. Anderson Guidelines for AE Reporting.

### 7.0 References

- 1. Oyen, RH, Van Poppel HP, Ameye FE, et al. Lymph node staging of localized prostatic carcinoma with CT and CT-guided fine-needle aspiration biopsy: prospective study of 285 patients. Radiology 1994; 190:315-322.
- 2. Dooms GC, Hricak H, Crooks LE, et al. Magnetic resonance imaging of the lymph nodes: comparison cith CT. Radiology 1984; 153:719-728.
- 3. Lee JK, Heiken JP, Ling D, et al. Magnetic resonance imaging of abdominal and pelvic lymphadenopathy. Radiology 1984; 153:181-188
- 4. Kim SH, Kim SC, Choi BI, et al. Uterine cervical carcinoma: evaluation of pelvic lymph node metastasis with MR imaging. Radiology 1994; 190:807-811.
- 5. Jager GJ, Barentsz JO, Oosterhof GO, et al. Pelvic adenopathy in prostatic and urinary bladder carcinoma: MR imaging with a three-dimensional T1-weighted magnetization-prepared-rapid gradient-echo sequence. AJR Am J Roentgenol 1996; 167:1503-1507.
- 6. Johnson JT. A surgeon looks at cervical lymph nodes. Radiology 1990; 175:607-610.
- 7. Ali S, Tiwari RM, Snow GB. False-positive and false-negative neck nodes. Head Neck Surg 1985; 8:78-82.
- 8. Guimaraes AR, Tabatabei S, Dahl D, et al. Pilot study evaluating use of lymphotrophic nanoparticle-enhanced magnetic resonance imaging for assessing lymph nodes in renal cell cancer. Urology 2008;71(4):708-712.
- 9. Tokuhara T, Tanigawa N, Matsuki M, et al. Evaluation of lymph node

Metastases in gastric cancer using magnetic resonance imaging with ultrasmall superparamagnetic iron oxide (USPIO): diagnostic performance in post-contrast images using new diagnostic criteria. Gastric Cancer 2008; 11(4):194-200.

10. Baghi M, Mack MG, Wagenblast J, et al. Iron oxide particle-enhanced magnetic resonance imaging for detection of benign lymph nodes in the head and neck: how reliable are the results? Anticancer research 2007; 27(5B):3571-3575.

- 11. Koh DM, Brown G, Temple L, et al. Rectal cancer: mesorectal lymph nodes at MR imaging with USPIO versus histopathologic findings--initial observations. Radiology 2004;231(1):91-99.
- 12. Rockall AG, Sohaib SA, Harisinghani MG,et. al. Diagnostic performance of nanoparticle-enhanced magnetic resonance imaging in the diagnosis of lymph node metastases in patients with endometrial and cervical cancer. J Clin Oncol 2005;23(12):2813-2821
- 13. Sigal R, Vogl T, Casselman J, et al. Lymph node metastases from head and neck
- squamous cell carcinoma: MR imaging with ultrasmall superparamagnetic iron oxide particles (Sinerem MR) results of a phase-III muticenter clinical trial. Eur Radiol 2002; 12:1104-1113.
- 14. Harisinghani MG, Barentsz J, Hahn PF, et al. Noninvasive detection of clinically occult lymph-node metastases in prostate cancer. N Engl J Med 2003; 348:2491-2499.
- 15. Feraheme®Package Insert http://www.amagpharma.com/documents/feraheme productinsert.pdf
- 16. Advanced Magnetics I. Magnetic Resonance Contrast Enhancement Agent
  - (Investigator's Drug Brochure). In. Cambridge, MA: Advanced Magnetics, Inc., 2002; 1-24.
- 17. Jung CW, Jacobs P. Physical and chemical properties of superparamagnetic iron oxide MR contrast agents: ferumoxides, ferumoxtran, ferumoxsil. Magn Reson Imaging 1995; 13:661-674.
- 18. Chambon C, Clement O, Le Blanche A, et al.. Superparamagnetic iron oxides a
- positive MR contrast agents: in vitro and in vivo evidence. Magn Reson Imaging 1993; 11:509-519.
- 19. Harisinghani MG, Barentsz J, Hahn PF, et al. Noninvasive detection of clinical
- occult lymph-node metastases in prostate cancer. N Engl J Med 2003; 348:2491-2499
- 20. Mayo-Smith WW, Saini S, Slater G, et al.. MR contrast material for vascular
- enhancement: value of superparamagnetic iron oxide. AJR 1996; 166(1):73-77 21. Reimer P, Muller M, Marx C, et al., T1 Effects of a Bolus-injectable Superparamagnetic
- Iron Oxide, SU U 555 A: Dependence on Field Strength and Plasma Concentration -
- Preliminary Clinical Experience with Dynamic T1-weigheted MR Imaging. Radiol 1998;
- 209; 831-836.